CLINICAL TRIAL: NCT01331525
Title: A Phase II Trial of the Addition of Ipilimumab to Carboplatin and Etoposide Chemotherapy for the First Line Treatment of Extensive Stage Small Cell Lung Cancer (ICE)
Brief Title: The Addition of Ipilimumab to Carboplatin and Etoposide Chemotherapy for Extensive Stage Small Cell Lung Cancer
Acronym: ICE
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: University Hospital Southampton NHS Foundation Trust (Other)
Collaborators: Cancer Research UK (Other); Institute of Cancer Research, United Kingdom (Other); Bristol-Myers Squibb (Industry)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: RHM CAN0739
Record Dates: First submitted 2011-04-04; First posted 2011-04-08 (Estimated); Last update posted 2016-04-14 (Estimated); Status verified 2016-04

CONDITIONS: Extensive Stage Small Cell Lung Cancer
Keywords: Small cell lung cancer; Chemotherapy; Immunotherapy; CTLA-4; Ipilimumab
MeSH Terms: conditions — Small Cell Lung Carcinoma; Diabetes Mellitus, Insulin-Dependent, 12 | interventions — Ipilimumab

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (1):
- Single stage non-randomised (Experimental): Patients will receive Carboplatin and Etoposide. Both Chemotherapy drugs will be delivered as a 21 day cycle (q21) with up to a maximum of 6 cycles delivered according to response unless progressive disease (RECIST Version 1.0) and or excessive toxicity.
  Ipilimumab will be administered at a dose of 10mg/kg IV on day 1 of cycles 3-6 of Chemotherapy.
  In the absence of immune related progression of disease or unacceptable toxicity, subsequent maintenance doses of Ipilimumab will be delivered every 12 weeks starting at week 30 at a dose of 10 mg/kg until unacceptable toxicity or immune related disease progression
  Interventions: Biological: Ipilimumab

INTERVENTIONS:
Biological: Ipilimumab — This trial will investigate the addition of the anti-CTLA4 antibody ipilimumab to conventional carboplatin and etoposide chemotherapy in extensive stage small cell lung cancer.
  Other Names: Yervoy; MDX-010; BMS-734016

SUMMARY:
This trial will investigate the addition of an antibody (Ipilimumab) to conventional Carboplatin and Etoposide chemotherapy in extensive stage small cell lung cancer.

The primary objective is to establish the progression free survival at 1 year.

DETAILED DESCRIPTION:
A Phase II trial of the addition of Ipilimumab to Carboplatin and Etoposide chemotherapy for the first line treatment of extensive stage small cell lung cancer (ICE)

Indication:

Extensive Stage Small cell lung cancer

Primary Objective:

To establish the progression free survival at 1 year in patients with extensive stage small cell lung cancer treated with ipilimumab, carboplatin and etoposide.

Secondary Objective:

To assess the response to and toxicity of the combination of ipilimumab with carboplatin and etoposide chemotherapy.

Immunological Objectives:

1. To examine whether ipilimumab stimulates a humoral immune response to onco-neuronal self-antigens

   The results from the above measurement of antibodies against onco-neuronal antigens will be used to focus the cellular biomarker analysis and identify targets to assess cellular responses:
2. To measure the effect of ipilimumab on CD8+ T-cells directed against onco-neuronal antigens, presumed to be responsible for the desired cytotoxic activity against cancer cells.
3. To evaluate the immune response to non-neuronal antigens in the presence of ipilimumab.

Rationale:

Small cell lung cancer accounts for around 20% of all lung cancer presentation in the UK. Of these approximately half present with extensive disease, overall representing 4000 new cases annually. Although initial response to chemotherapy for this group of patients ranges from 50-60% 1, 2, subsequent relapse is inevitable and results in poor survival with only 5% of patients alive at 2 years from diagnosis.

Despite attempts to improve on conventional chemotherapy with platinum and etoposide in extensive stage small cell lung cancer, neither modification of conventional chemotherapeutic drugs, nor the use of novel targeted therapy has shown an increased benefit. A conceptual change in therapeutic strategy is therefore required, and immunotherapy is an attractive avenue to pursue.

Anti-CTLA4 antibody may allow the development or induction of anti-tumour immunity even in the absence of a known tumour antigen and without active anti-tumour vaccination. Chemotherapy effectively kills tumour cells and releases tumour derived antigens and as such administration of anti-CTL4 antibody may induce a clinically useful anti-tumour immune response against these antigens.

This trial will therefore investigate the addition of the anti-CTLA4 antibody ipilimumab to conventional carboplatin and etoposide chemotherapy in extensive stage small cell lung cancer.

Trial Design:

Single stage non-randomised phase II trial

Sample size:

Patients will be recruited so that 40 patients are treated with chemo-immunotherapy. If 8 or more patients are progression free at 1 year the treatment will be considered to be successful and warrant further testing.

Study Population:

All patients consented will form the ITT population.

• Patients who have received at least 1 dose of Ipilimumab will form the analysis population (N=40).

Dosage Regimen/Duration of Treatment:

Subjects will receive up to 6 cycles of carboplatin and etoposide chemotherapy according to response and toxicity. Carboplatin will be administered at a dose of AUC = 6 (calculated according to the Calvert formula using a Cockcroft and Gault calculation of creatinine clearance) IV, day 1.

Etoposide will be administered at 120mg/m2 IV day 1, 100mg BD PO days 2 and 3. Both chemotherapy drugs will be delivered as a 21 day cycle (q21) with up to a maximum of 6 cycles delivered according to response unless progressive disease (RECIST) and or excessive toxicity.

Ipilimumab will be administered at a dose of 10mg/kg IV on day 1 of cycles 3-6 of chemotherapy.

In the absence of immune related progression of disease or unacceptable toxicity, subsequent maintenance doses of ipilimumab will be delivered every 12 weeks starting at week 30 at a dose of 10 mg/kg until unacceptable toxicity or immune related disease progression.

Tumour assessments:

Tumour assessments by CT scanning of the chest, abdomen and pelvis will be performed at baseline and the following time points until progression:

Weeks 6, 12, 18, 24, 30, 36, 42, 48, 52 and then 12 weekly until progression by both RECIST and immune related response criteria.

Duration of study:

It is expected that with the current standard of care the trial will take 24 months to recruit with completion of the trial anticipated in 3 years. The study may however continue for longer if patients are continuing to receive maintenance ipilimumab, in which case the study will finish 100 days after the last dose of ipilimumab (when it is clear the last dose has been given) or when all patients have died.

Safety monitoring:

Given the different safety profile of ipilimumab and carboplatin / etoposide chemotherapy, no overlapping toxicity is expected.

However, throughout the trial, there will be a close monitoring of the nature and the severity of the adverse events reported on an on-going basis.

A planned interim safety monitoring assessment will be performed. Once 9 patients have been treated with the combination for at least 6 weeks (subjects who discontinued treatment earlier due to excessive toxicity of chemo-immunotherapy will also be considered), a first clinical safety assessment will be performed to identify any early safety signals from ipilimumab given in combination with carboplatin and etoposide.

In addition a review of safety may be triggered throughout the trial:

If greater than or equal to 40% of subjects treated develop a greater than or equal to Grade 3 toxicity thought to be related to the study drugs; or If greater than or equal to 10% of subjects experience an unexpected ipilimumab-related greater than or equal to Grade 3 toxicity that cannot be alleviated or controlled by appropriate care and/or steroid and/or infliximab therapy within 14 days of the initiation of such therapy.

In response to any ipilimumab-related deaths unless attributed to disease progression.

In these circumstances the data will be carefully reviewed to determine the appropriate course of action, which could include:

Continue without modification; Continue with modifications of the study protocol. Modifications may include, but are not limited to, changes in inclusion/exclusion criteria, frequency of safety monitoring, change in ipilimumab dose, and alterations in study procedures; Discontinue the study (with provisions for orderly discontinuation in accordance with good medical practice) under extreme circumstances (eg, insufficient benefit-to-risk effect of the experimental treatment).

The decision to put patient accrual on hold while reviewing safety data will be taken or not, based on characteristics of the serious adverse events reported on an ongoing basis.

The review will take into account the known toxicity profile for ipilimumab and for carboplatin/etoposide, and the potential association of immune-related Adverse Events (irAEs) with clinical efficacy.

ELIGIBILITY:
Inclusion Criteria:

* Willing and able to give written informed consent.
* Histological or cytological diagnosis of small cell lung cancer.
* Adequate baseline laboratory tests.
* No active or chronic infection with HIV, Hepatitis B, or Hepatitis C.
* Performance status ECOG 0 or 1.
* Men and women, 18 years of age and above.

Exclusion Criteria:

* Limited stage small cell lung cancer appropriate for radical treatment with chemoradiation.
* Symptomatic CNS metastases.
* A history of prior malignant tumour, unless the patient has been without evidence of disease for at least 5 years, with the exception of adequately treated basal or squamous cell skin cancer, superficial bladder cancer or carcinoma in situ of the cervix.
* Clinically significant autoimmune disease.
* Any underlying medical, neurological or psychiatric condition, which in the opinion of the investigator will make the administration of ipilimumab hazardous or obscure the interpretation of AEs.
* Administration of any live vaccine for prevention of infectious diseases (for up to 1 month before or after any dose of ipilimumab).
* Previous chemotherapy for small cell lung cancer.
* A history of prior treatment with immunostimulatory antibodies ipilimumab, prior CD137 agonist or CTLA 4 inhibitor or agonist.
* Concomitant therapy with any of the following: Interleukin 2, interferon, or other non-study immunotherapy regimens; immunosuppressive agents; other investigation therapies; or chronic use of systemic corticosteroids.
* Women of childbearing potential (WOCBP), as defined in the protocol and who:

  * Are unwilling or unable to use an acceptable method of contraception to avoid pregnancy for the duration of their participation in the study and for at least 8 weeks after cessation of study drug, or
  * Have a positive pregnancy test at baseline, or
  * Are pregnant or breastfeeding.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 42 (Actual)
Dates: Start 2011-06; Primary Completion 2015-06 (Actual); Study Completion 2015-06 (Actual)

PRIMARY OUTCOMES:
To establish the progression free survival at 1 year in patients with extensive stage small cell lung cancer treated with ipilimumab, carboplatin and etoposide. | At 1 year from entering trial

SECONDARY OUTCOMES:
Assess tumour response and toxicity of ICE combination. Response measured by RECIST and immune related response criteria. Toxicity via physical exam, adverse event review, assessing signs and symptoms, quality of life assessment and blood testing. | Throughout clinical trial participation (maximum 6 21 day cycles) plus 100 day follow up from last treatment.
  Response: Assessed via Chest X-ray and CT of chest, abdomen and pelvis at weeks 6, 12, 18, 24, 30, 36, 42, 48, 52 and then 12 weekly until progression.
  Toxicity: targeted physical, adverse event assessment, assessment of signs and symptoms, quality of life assessment, full blood count plus ALT/ASP, ALP, Billi, Ca, Alb, LDH, Creatinine, urea and electrolytes investigation. Serious adverse events will be reported within 24 hours of first knowledge of the event.

CONTACTS AND LOCATIONS:
Overall Officials: Christian H Ottensmeier, MD, PhD, Study Chair — University Hospital Southampton NHS Foundation Trust; Matthew Wheater, MD, Principal Investigator — University Hospital Southampton NHS Foundation Trust
Locations (7):
- United Kingdom (7):
  - Royal Bournemouth Hospital, Bournemouth
  - Leeds Teaching Hospitals NHS Foundation Trust, Leeds
  - Barts and The London NHS Trust, London
  - The Clatterbridge Cancer Centre NHS Foundation Trust, Metropolitan Borough of Wirral
  - Nottingham University Hospitals NHS Trust, Nottingham
  - Weston Park Clinical Trials Centre, Sheffield
  - Southampton University Hospitals NHS Trust, Southampton

IPD SHARING:
Plan to Share IPD: Yes